CLINICAL TRIAL: NCT00744380
Title: Dexmedetomidine vs. Midazolam for Facilitating Extubation in Medical and Surgical ICU Patients: A Randomized, Double-Blind Study
Brief Title: Dexmedetomidine Versus Midazolam for Facilitating Extubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-0570
Record Dates: First submitted 2008-08-28; First posted 2008-09-01 (Estimated); Results first posted 2016-09-28 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-08

CONDITIONS: Critical Illness
Keywords: Analgesia; Mechanical ventilation
MeSH Terms: conditions — Critical Illness; Agnosia | interventions — Midazolam; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Midazolam (Active Comparator): Midazolam infusion of 1 mg/hour (final infusion concentration of 0.5 mg/mL) and adjusted by 1 mg/hour by the bedside nurse as needed for the desired level of sedation (Riker sedation-agitation score of 3 - 4) as other sedatives are down titrated. Daily awakenings are used.
  Interventions: Drug: Midazolam
- Dexmedetomidine (Experimental): Dexmedetomidine 0.15 µg/kg per hour (final infusion concentration of 0.075 µg/kg per mL) and adjusted by 0.15 µg/kg per hour by the bedside nurse as needed for the desired level of sedation (Riker sedation-agitation score of 3 - 4)as other sedatives are down titrated. Daily awakenings are used.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Midazolam — Midazolam infusion of 1 mg/hour (final infusion concentration of 0.5 mg/mL) and adjusted by 1 mg/hour by the bedside nurse as needed for the desired level of sedation (Riker sedation-agitation score of 3 - 4)
  Other Names: Versed
  Arms: Midazolam
Drug: Dexmedetomidine — Dexmedetomidine 0.15 µg/kg per hour (final infusion concentration of 0.075 µg/kg per mL) and adjusted by 0.15 µg/kg per hour by the bedside nurse as needed for the desired level of sedation (Riker sedation-agitation score of 3 - 4)
  Other Names: Precedex
  Arms: Dexmedetomidine

SUMMARY:
The purpose of this randomized, double-blind study is to evaluate the utility, safety, and cost of transitioning benzodiazepine sedation to dexmedetomidine in medical or surgical intensive care unit (ICU) patients requiring sedation when tracheal extubation is nearing. Fifty medical or surgical ICU patients requiring sedation with existing benzodiazepine therapy and qualifying for daily awakenings will be randomized in a double-blind manner to receive additional midazolam or dexmedetomidine.

DETAILED DESCRIPTION:
This study is unique because midazolam or dexmedetomidine will be added, in a blinded fashion, to existing sedation and analgesia in an effort to decrease or possibly discontinue these therapies.

Objectives:

The objectives of this study are to determine if transitioning conventional sedation to dexmedetomidine safely facilitates tracheal extubation after study initiation; alters the amounts of sedative and analgesic agents required after study initiation; influences the levels of sedation and analgesia; alters the adverse event profile (neurologic, hemodynamic, or gastrointestinal) during and after discontinuing sedation; and impacts the total cost of sedation during and after discontinuing sedation.

Hypothesis 1: Transitioning conventional sedation to dexmedetomidine expedites tracheal extubation to shorten ventilator time.

Specific Aim 1: Comparatively determine the time from study initiation to tracheal extubation with midazolam and dexmedetomidine when the practice of daily awakenings is used.

Hypothesis 2: Transitioning conventional sedation to dexmedetomidine reduces the doses of conventional sedatives and analgesics while maintaining equivalent levels of sedation and analgesia and not incurring adverse events.

Specific Aim 2a: Comparatively determine the hourly, daily, and cumulative doses of conventional sedatives and analgesics from study initiation to sedation discontinuation with midazolam and dexmedetomidine when the practice of daily awakenings is used.

Specific Aim 2b: Comparatively evaluate the quality of sedation and analgesia of midazolam and dexmedetomidine by determining the proportion of Riker sedation scores at 3 - 4 (desired level of sedation) and ≤ 2 or ≥ 5 (undesired levels of sedation) and the proportion of Pain Assessment Behavioral Scores (PABS) ≤ 3 (comfortable) and ≥ 4 (pain).

Specific Aim 2c: Comparatively evaluate sedation-related adverse effects (neurologic, hemodynamic, or gastrointestinal) of midazolam and dexmedetomidine when the practice of daily awakenings is used.

Hypothesis 3: Transitioning conventional sedation to dexmedetomidine increases the cost of administering sedation but minimizes the incidental costs associated with sedation to counterbalance and possibly reduce the total cost of sedation (sum of administration costs and incidental costs).

Specific Aim 3a: Comparatively determine the hourly, daily, and cumulative administration costs of midazolam and dexmedetomidine when the practice of daily awakenings is used.

Specific Aim 3b: Comparatively determine the hourly, daily, and cumulative incidental costs of conventional sedatives and dexmedetomidine; including neurologic dysfunction, antipsychotic requirements, cardiovascular dysfunction, constipation or ileus, differences in times to ventilator discontinuation, personnel time, and patient transfer from the ICU after sedation discontinuation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients requiring mechanical ventilation in the medical or surgical ICUs.
2. Currently receiving lorazepam or midazolam by continuous infusion for the purpose of sedation therapy.
3. Sedation in these ICUs is provided using an ICU-wide order form that preferentially uses either lorazepam or midazolam with the infusion rate titrated by the bedside nurse to the desired Riker sedation-agitation score(s). Continuous analgesia is provided with fentanyl only with the infusion rate titrated by the bedside nurse to PABS ≤ 3 .
4. Anticipated duration of continuous sedation > 12 hours with the level of sedation expected to be maintained at Riker sedation-agitation score(s) of 3 - 4.
5. Patients qualifying for daily awakenings as determined by all of the following:

   * fraction of inspired oxygen (FiO2) ≤ 70% or
   * positive end expiratory pressure (PEEP) ≤ 14 cmH2O,
   * hemodynamically stable, and
   * NOT receiving pharmacologic neuromuscular blockade.
6. Informed consent and HIPAA authorization within 24 hours of qualifying for daily awakenings.

Exclusion Criteria:

1. Patients < 18 years of age or > 85 years of age.
2. Patients receiving intermittent or "as needed" administration of lorazepam or midazolam.
3. Patients receiving lorazepam or midazolam for purposes other than sedation (e.g. seizure control).
4. Patients receiving epidural administration of medication(s).
5. Patients with Childs-Pugh class C liver disease.
6. Comatose patients by metabolic or neurologic affectation.
7. Patients with active myocardial ischemia or second- or third-degree heart block.
8. Moribund state with planned withdrawal of life support.
9. Patients with known or suspected severe adverse reactions to midazolam (or any other benzodiazepine) or dexmedetomidine (or clonidine).
10. Patients with alcohol abuse within six months of study eligibility.
11. Pregnant females or females suspected of being pregnant.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert MacLaren, PharmD, Principal Investigator — University of Colorado Skaggs School of Pharmacy and Pharmaceutical Sciences
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Publication

REFERENCES:
- [Derived] MacLaren R, Preslaski CR, Mueller SW, Kiser TH, Fish DN, Lavelle JC, Malkoski SP. A randomized, double-blind pilot study of dexmedetomidine versus midazolam for intensive care unit sedation: patient recall of their experiences and short-term psychological outcomes. J Intensive Care Med. 2015 Mar;30(3):167-75. doi: 10.1177/0885066613510874. Epub 2013 Nov 12. PMID 24227448

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Midazolam | Dexmedetomidine
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Midazolam | Dexmedetomidine | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (9.3) | 58.3 (15.3) | 58.1 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 7 | 6 | 13
Weight [Mean (Standard Deviation); unit: kg] | 105.2 (40.9) | 100.8 (37.4) | 103 (38.5)
Acute Physiologic And Chronic Health Evaluation III Score [Mean (Standard Deviation); unit: units on a scale] — APACHE III measures the severity of disease for adult patients admitted to intensive care units. The point score is calculated as a summation from scores assigned to a patient's age, primary comorbidity, preexisting comorbidities, location prior to ICU admission, Glasgow Coma Scale, and 20 routine physiological measurements. APACHE III scores range from 0 to 299. This provides an initial risk classification of severely ill hospitalized patients in defined groups with higher scores indicating greater disease severity and correlated to higher mortality risk.
  units on a scale | 70.4 (33.5) | 74.1 (18.2) | 72.8 (25)
Primary Diagnosis [Number; unit: participants]
  Respiratory failure | 5 | 5 | 10
  Sepsis | 5 | 4 | 9
  Other | 2 | 2 | 4
Time in ICU before qualifying [Median (Inter-Quartile Range); unit: days] | 1.1 [0.6 to 2] | 1.2 [0.9 to 5.4] | 1.1 [0.6 to 5.4]
Time from qualifying to randomization [Median (Inter-Quartile Range); unit: days] | 1 [0.7 to 1.1] | 0.7 [0.5 to 0.8] | 0.9 [0.5 to 1.1]
Baseline Sedative [Number; unit: participants]
  Midazolam | 10 | 6 | 16
  Lorazepam | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Time From Study Drug Initiation to Tracheal Extubation
Time Frame: Duration of ICU stay, for up to 24 weeks
Population: The analysis only includes patients successfully extubated for at least 72 hours. Eight subjects were excluded.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Midazolam | Dexmedetomidine
Number analyzed (Participants) | 8 | 7
days | 2.9 [2 to 4.4] | 3.4 [2.6 to 14.2]
Statistical Analysis 1: Comparison: Midazolam vs Dexmedetomidine; Test type: Superiority or Other; p = 0.8, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Cumulative Doses of Conventional Sedatives and Analgesics
Time Frame: Duration of ICU stay, for up to 24 weeks
Measure: Median (Inter-Quartile Range); unit: mg
Groups:
- Dexmedetomidine: Dexmedetomidine 0.15 µg/kg per hour (final infusion concentration of 0.075 µg/kg per mL) and adjusted by 0.15 µg/kg per hour by the bedside nurse as needed for the desired level of sedation (Riker sedation-agitation score of 3 - 4) as other sedatives are down titrated. Daily awakenings are used.
  Dexmedetomidine: Dexmedetomidine 0.15 µg/kg per hour (final infusion concentration of 0.075 µg/kg per mL) and adjusted by 0.15 µg/kg per hour by the bedside nurse as needed for the desired level of sedation (Riker sedation-agitation score of 3 - 4)
Arm/Group | Midazolam | Dexmedetomidine
Number analyzed (Participants) | 12 | 11
mg
  Open-label midazolam while on study drug | 29 [18.8 to 48.9] | 65.3 [24.5 to 92.3]
  All midazolam whil eon study drug | 126.9 [93.2 to 608.8] | 65.3 [24.5 to 92.3]
  All fentanyl while on study drug | 5.4 [3.5 to 9.2] | 4.1 [3 to 14]
Statistical Analysis 1: Comparison: Midazolam vs Dexmedetomidine; For open label midazolam; Test type: Superiority or Other; p = 0.25, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Midazolam vs Dexmedetomidine; For all midazolam; Test type: Superiority or Other; p = 0.048, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Midazolam vs Dexmedetomidine; For fentanyl; Test type: Superiority or Other; p = 0.88, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: The Quality of Sedation (Assessed by the Riker Sedation-Agitation Score) and Analgesia (Assessed by the Pain Assessment Behavioral Score)
Description: The Riker sedation-agitation score (range 1-7) and PABS (range 0-10) are assessed hourly by the bedside nurse. Riker scores assess restlessness and cooperation. Riker scores of 5 - 7 indicate agitation, 3 - 4 represent adequate sedation and 1 - 2 represent excessive sedation. PABS assessments include domains of restlessness, muscle tone, vocalization, consolability, and facial expressions. PABS assessments of 0 represent no pain, 1 - 3 represent mild pain, 4 - 6 represent moderate pain, and ≥ 7 represent severe pain.
Time Frame: Duration of ICU stay, for up to 24 weeks
Measure: Number; unit: percentage of assessments while on study
Arm/Group | Midazolam | Dexmedetomidine
Number analyzed (Participants) | 12 | 11
percentage of assessments while on study
  Riker score 1-2 while on study drug | 5.4 | 4.1
  Riker score 3-4 while on study drug | 84.1 | 71.2
  Riker score 5-7 while on study drug | 6.6 | 27.1
  Pain score > 3 while on study drug | 13.3 | 21.4
Statistical Analysis 1: Comparison: Midazolam vs Dexmedetomidine; For Riker scores; Test type: Superiority or Other; p = 0.75, Chi-squared, Corrected
Statistical Analysis 2: Comparison: Midazolam vs Dexmedetomidine; For pain scores; Test type: Superiority or Other; p = 0.17, Chi-squared

4. Secondary Outcome: Sedation-related Adverse Effects
Time Frame: Duration of ICU stay, up to 24 weeks
Measure: Number; unit: participants
Arm/Group | Midazolam | Dexmedetomidine
Number analyzed (Participants) | 12 | 11
participants
  Hypotension | 6 | 10
  Bradycardia | 7 | 7
  Tachycardia | 5 | 7
  Delirium, new onset | 5 | 1
Statistical Analysis 1: Comparison: Midazolam vs Dexmedetomidine; For hypotension; Test type: Superiority or Other; p > 0.1, Chi-squared, Corrected
Statistical Analysis 2: Comparison: Midazolam vs Dexmedetomidine; For bradycardia; Test type: Superiority or Other; p > 0.1, Chi-squared, Corrected
Statistical Analysis 3: Comparison: Midazolam vs Dexmedetomidine; For tachycardia; Test type: Superiority or Other; p > 0.1, Fisher Exact
Statistical Analysis 4: Comparison: Midazolam vs Dexmedetomidine; For delirium, new onset; Test type: Superiority or Other; p = 0.07, Fisher Exact

5. Secondary Outcome: ICU Experiences by Administering ICU Stressful Experiences Questionnaire (ICU-SEQ)
Description: The ICU-SEQ assesses patient recall of their ICU experience. The ICU-SEQ assesses both psychological (e.g. fearfulness, anxiety) and physical (e.g. pain, difficulty breathing) perceptions of ICU patients who have received mechanical ventilation. It consists of 29 potentially stressful experiences with seven items specifically addressing the endotracheal tube. The extent that patients are bothered by each item is scored on a five point scale: 0 = "not at all," 1 = "a little bit," 2 = "moderately," 3 = "quite a bit," and 4 = "extremely." The cumulative score is an integer interpreted as interval data with higher scores indicating greater stressful experiences associated with the ICU. The minimum score is 0 and the maximum score possible is 116.
Time Frame: Duration of hospital stay, up to 24 weeks
Population: Only subjects capable of performing the ICU-SEQ were provided the assessment. Seven subjects were excluded.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Midazolam | Dexmedetomidine
Number analyzed (Participants) | 8 | 8
units on a scale | 8.5 [0 to 29] | 18.5 [0 to 29]
Statistical Analysis 1: Comparison: Midazolam vs Dexmedetomidine; Median number of experiences remembered; Test type: Superiority or Other; p = 0.015, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Duration of Study Drug Administration
Time Frame: Duration of ICU stay, up to 24 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Midazolam | Dexmedetomidine
Number analyzed (Participants) | 12 | 11
days | 3 [0.8 to 5.1] | 3.5 [2 to 4.9]
Statistical Analysis 1: Comparison: Midazolam vs Dexmedetomidine; Test type: Superiority or Other; p = 0.5, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Manifestations of Acute Stress Disorder by Impact of Event Scale - Revised (IES-R)
Description: The IES-R evaluates subjective distress caused by traumatic events and assesses manifestations of post-traumatic stress disorder (PTSD) or acute stress disorder. It is not diagnostic but possesses excellent reliability and validity for manifestations of PTSD. The IES-R has three subscales (eight items on intrusion, eight items on avoidance, and six items on hyperarousal). Each item is scored on a four point scale: 0 = "not at all," 1 = "a little bit," 2 = "moderately often," 3 = "quite a bit," and 4 = "extremely often." The total score of each subscale may be averaged and a cumulative score of 30 is indicative of the presence of PTSD. The maximum score for each subscale is 32 for intrusion, 32 for avoidance, and 24 for hyperarousal. The minimum cumulative score is 0 and the maximum cumulative score possible is 88.
Time Frame: Duration of hospital stay, up to 24 weeks
Population: Only subjects capable of performing the IES-R were provided the assessment. Seven subjects were excluded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Midazolam | Dexmedetomidine
Number analyzed (Participants) | 8 | 8
units on a scale | 13 (12) | 36 (12)
Statistical Analysis 1: Comparison: Midazolam vs Dexmedetomidine; Test type: Superiority or Other; p = 0.029, t-test, 2 sided

8. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) Score
Description: The HADS consists of 14 questions, seven for anxiety and seven for depression. Each item is scored from 0 to 3, with a cut-off cumulative score of 11 for both subscales indicative of anxiety or depression. This scoring tool has been used for 30 years, possesses excellent reliability and validity, and avoids reliance conditions that are also common somatic symptoms of illness such fatigue, insomnia, and hypersomnia. The maximum score for each subscale is 21 with a maximum possible cumulative score of 42. The minimum score for each subscale is 0. The minimum cumulative score is 0
Time Frame: Duration of hospital stay, up to 24 weeks
Population: Only subjects capable of performing the HADS were provided the assessment. Seven subjects were excluded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Midazolam | Dexmedetomidine
Number analyzed (Participants) | 8 | 8
units on a scale
  Anxiety | 3 (3.1) | 6 (7.6)
  Depression | 6 (6.7) | 4 (5.3)
Statistical Analysis 1: Comparison: Midazolam vs Dexmedetomidine; For anxiety; Test type: Superiority or Other; p > 0.1, t-test, 2 sided
Statistical Analysis 2: Comparison: Midazolam vs Dexmedetomidine; For depression; Test type: Superiority or Other; p > 0.1, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Midazolam | Dexmedetomidine
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/11
Other Adverse Events (participants affected / at risk) | 12/12 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Midazolam (N=12) | Dexmedetomidine (N=11)
Acute Neurologic Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Midazolam (N=12) | Dexmedetomidine (N=11)
Hypotension (Cardiac disorders) | 6 (6) | 10 (10)
Bradycardia (Cardiac disorders) | 7 (7) | 7 (7)
Tachycardia (Cardiac disorders) | 5 (5) | 7 (7)
Delirium, new onset (Nervous system disorders) | 5 (5) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes